CLINICAL TRIAL: NCT05461443
Title: Study of the Modularity Immune Function of Lactobacillus Rhamnosus GG in the Small Intestine of Healthy Individuals
Brief Title: Lacticaseibacillus Rhamnosus GG Pili Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Valio Ltd (Industry); Chr Hansen (Industry)
Responsible Party: Principal Investigator, Robert Brummer, Professor, Örebro University, Sweden
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015/422
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Lacticaseibacillus rhamnosus GG; Probiotics; Pili; Gut microbiota; Transcriptomics; Small intestine
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The individuals did receive the three treatment combinations in a randomised order.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The sachets containing the different LGG strains were labelled as A, B, and C. The codes for each strain were kept by the industrial partner that provided the probiotic strains. Only at the end of the data analyses were the codes disclosed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Wild-type (Active Comparator): Supplementation with the wild-type of the LGG strain
  Interventions: Dietary Supplement: Probiotic
- Low-pill (Experimental): Supplementation with the low-pili LGG strain
  Interventions: Dietary Supplement: Probiotic
- High-pili (Experimental): Supplementation with the high-pili LGG strain
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic
  Other Names: LGG

SUMMARY:
The aim of this study was to investigate the host-microbe interaction effects of various Lacticaseibacillus rhamnosus GG strains, with different binding capacities to the mucus in the small intestine, in healthy individuals

DETAILED DESCRIPTION:
The project consisted in the supplementation of a) a wild-type LGG strain, b) a low-producing pili LGG strain or c) a high-producing pili LGG strain to study subjects. The individuals received the three treatment combinations in a randomised order. Each supplementation was given to the individuals every 30 min over a period of 6 hours. Eight biopsies from the duodenum were collected at the end of 6 h-solutions administration by flexible gastroduodenoscopy, likewise the routine procedure during this endoscopic investigation. Faecal samples were collected by the study subjects at home 1 day before, 2, 7 and 14 days days after administrations of each oral supplementation. The supplementations were separated by a 3-week wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-65 years.
* Willing to abstain from any probiotics or medication known to alter gastrointestinal function during the study.
* A signed informed consent.

Exclusion Criteria:

* Recent or current treatment with drugs affecting intestinal function, immune function or mood (e.g. antidepressants). In addition use of all drugs during the study should be recorded.
* Recent (< 6 weeks) use of probiotics*.
* Diagnosis of major psychiatric or somatic disorders.
* Pregnancy or breastfeeding.
* Abuse of alcohol or drugs.
* Smokers and chewable tobacco users.
* Lactose intolerance.

  * Any kind of probiotics and with special attention on products containing LGG:

Dairy products:

* Valio Kefir
* Valio Gefilus yoghurt

Dietary supplements:

* Bifiform Daily
* Bifiform Travel
* Bifiform Daily Caps

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in whole genome gene expression of duodenal mucosa after administration of three different LGG strain | 6hrs supplementation after start of LGG strain administration.
  Microarray-based Gene expression Analysis were carried out from duodenal biopsies collected after the supplementation of each LGG strain
Microbiome of duodenal mucosal biopsies | 6hrs supplementation after start of LGG strain administration
  Bacterial composition was analysed by Illumina MiSeq sequencing the hypervariable V3-V4 region of the 16S rRNA gene

SECONDARY OUTCOMES:
Faecal microbiome | 2 days after LGG strain administration
  Bacterial composition by MiSeq sequencing hypervariable V3-V4 region of 16SrRNA gene
Faecal microbiome | 7 days after LGG strain administration
  Bacterial composition by MiSeq sequencing hypervariable V3-V4 region of 16SrRNA gene
Faecal microbiome | 14 days after LGG strain administration
  Bacterial composition by MiSeq sequencing hypervariable V3-V4 region of 16SrRNA gene

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, Professor, Study Director — Örebro University, School of Medical Sciences, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No